CLINICAL TRIAL: NCT00474084
Title: First In Man Evaluation of the Vesta™ & VestaCOR™ (Hydroxy-Apetite Coated genX™) Stent for Treatment of de Novo Native Coronary Artery Lesion(s)
Brief Title: Hydroxyapatite Active Pro Healing Clinical Trial Program
Acronym: HApFIM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: BioSync Scientific Pvt. Ltd. (Industry)
Collaborators: MIV Therapeutics Inc. (Industry); Cardialysis BV (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HAP/CT/01
Record Dates: First submitted 2007-05-15; First posted 2007-05-16 (Estimated); Last update posted 2007-05-16 (Estimated); Status verified 2007-05

CONDITIONS: Coronary Artery Disease
Keywords: Stent; Hydroxyapatite; Coronary Artery Stenosis; Angioplasty
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Intravascular Coronary Stent

SUMMARY:
The purpose of this first feasibility study is to evaluate the performance of Vesta™ & VestaCOR™ (Hydroxy-Apetite coated GenX) stent in de novo native coronary artery lesions. This study will provide the longest follow-up experience available.

This is a randomized, double blind study conducted at three sites, two sites in India and one in The Netherlands. To be eligible, a patient will be required to have a de novo stenotic lesion of a length that could be covered by a single stent in a native coronary artery of diameter 3.0mm and 3.5mm. A total of at least 60 patients and a maximum of 70 patients will be treated with Vesta™ & VestaCOR™ stent. These patients will be randomized to either a smooth surface nanofilm coated stent (= VestaCOR™) (approx. 35 patients) or to a porous coated stent (= Vesta™) (approx. 35 patients).

All patients will be followed clinically at 30 days, 4 months, 9 months, 1, 2, 3, 4 and 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient is  18 years old
* Patient is eligible for percutaneous coronary intervention (PCI)
* Patient is an acceptable candidate for CABG
* Clinical evidence of ischemic heart disease and/or a positive territorial functional study. Documented stable angina pectoris ((Canadian Cardiovascular Society (CCS) Classification 1, 2, 3 or 4) or unstable angina pectoris with documented ischemia (Braunwald Class IB-C, IIB-C, or IIIB-C), or documented silent ischemia
* The target lesion is a single de novo coronary artery lesion with 50 and 100% stenosis in one of the major epicardial territories (LAD, LCX or RCA). A second target lesion in another major epicardial vessel could be treated and this second lesion should fit with inclusion/exclusion criteria and will receive the same type of stent.
* The target lesion must be covered by one study stent preferably with a margin of at least 4mm on each side of the lesion
* The target lesion length should be ≤ 11 mm
* The target reference vessel diameter must be  3.0mm and  3.5mm
* Patient or the patient's legal representative has been informed of the nature of the study and agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board/Ethics Committee of the respective clinical site

Exclusion Criteria:

* Female of childbearing potential
* Documented left ventricular ejection fraction (LVEF) 30%
* Evidence of an acute Q-wave or non-Q-wave myocardial infarction within 72 hours preceding the index procedure, unless the CK and CK-MB enzymes are less than twice the Upper Normal Limit
* Known allergies to the following: aspirin, clopidogrel bisulfate (Plavix®) or ticlopidine (Ticlid®), heparin, Stainless Steel , contrast agent (that cannot be adequately pre-medicated) or drugs similar to hydroxyapatite
* A platelet count 100,000 cells/mm3 or 700,000 cells/mm3 or a WBC 3,000 cells/mm3
* Acute or chronic renal dysfunction (creatinine 2.0 mg/dl or 150µmol/L)
* Total occlusion (TIMI 0 or 1 (one))
* Target vessel has evidence of thrombus or is excessively tortuous that makes it unsuitable for proper stent delivery and deployment;
* Previous bare metal stenting (less than 1 year) anywhere within the target vessel
* Previous drug-eluting stenting anywhere within the target vessel;
* The target lesion requires treatment with a device other than PTCA prior to stent placement (e.g. but not limited to, directional coronary atherectomy, excimer laser, rotational atherectomy, etc.)
* Significant (50%) stenosis proximal or distal to the target lesion that might require revascularization or impede run off;
* Heavily calcified lesion and/or calcified lesion which cannot be successfully predilated
* Target lesion is located in or supplied by an arterial or venous bypass graft
* Ostial target lesion
* Target lesion involves a side branch 2.0mm in diameter with an ostial disease
* Patient is currently participating in an investigational drug or device study
* Within 30 days prior procedure patient has undergone a previous coronary interventional procedure of any kind
* Within 60 days post-procedure patient requires planned interventional treatment of any non-target vessel. Planned intervention of the target vessel after the index procedure is not allowed
* Stroke or transient ischemic attack within the prior 6 months
* Unprotected Left Main (LM) coronary artery disease (stenosis >50%)
* In the investigator's opinion patient has a co-morbid condition(s) that could limit the patient's ability to participate in the study, compliance with follow-up requirements or impact the scientific integrity of the study
* Planned surgery within 6 months after index procedure
* Life expectancy less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2007-07

PRIMARY OUTCOMES:
In-stent late-loss at 4 and 12 months (as measured by QCA), defined as the difference between the post-procedure minimal lumen diameter (MLD) and the follow-up angiographic MLD | 4 & 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrick W Serruys, PhD, Principal Investigator — Erasmus MC Thoraxcentrum, The Netherlands